CLINICAL TRIAL: NCT00578916
Title: Pharmacokinetics and Metabolism of [14C] BMS-690514 in Healthy Male Subjects
Brief Title: Pharmacokinetics and Metabolism of Radiolabeled BMS-690514 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA187-003
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2008-07-31 (Estimated); Status verified 2008-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — BMS-690514

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: EVRI (BMS-690514)

INTERVENTIONS:
Drug: EVRI (BMS-690514) — Oral Solution, Oral, 200 mg, single dose followed by 10-12 day inpatient stay

SUMMARY:
The purpose of this study is to determine how the human body processes and eliminates the drug (BMS-690514.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Body mass index (BMS) of 18 - 30 kg/m², inclusive

Exclusion Criteria:

* Radiation exposure from diagnostic X-rays (except dental X-rays) in the last year or from clinical trials in the last 5 years

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2008-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Single dose pharmacokinetics of BMS-690514 and radioactivity in plasma and urine | measured for 10 days post-dose

SECONDARY OUTCOMES:
Determination of biotransformation profiles and recorded adverse events | for 10 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Allschwil, Switzerland